CLINICAL TRIAL: NCT04540952
Title: A Prospective, Randomized Trial to Compare the Fluid Capture Efficiency of the "Total Capture" Drape Versus a Standard Drape for Hysteroscopy: Innovation for Improved Patient Safety and Surgical Care.
Brief Title: Comparison of Fluid Capture Efficiency of the Total Capture Drape Versus a Standard Drape for Hysteroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: North Carolina Biotechnology Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 04-16-07B
Record Dates: First submitted 2020-06-29; First posted 2020-09-07 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-11

CONDITIONS: Hysteroscopic Surgery
Keywords: hysteroscopy; fluid management; safety; surgical complications; surgical drape

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Early Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomization of patients without their knowledge of grouping. Surgical providers become aware of randomized drape selection only at the time of hysteroscopy. Principal investigator blinded to selection and results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Total Capture Drape (Experimental): Surgical drape created by Principal Investigator to adequately collect fluid during hysteroscopy procedure
  Interventions: Device: Total Capture Drape
- Control (Active Comparator): Standard surgical drape used to adequately collect fluid during hysteroscopy procedure
  Interventions: Device: Standard Hysteroscopy Drape

INTERVENTIONS:
Device: Total Capture Drape — Surgical drape created by Principal Investigator to adequately collect fluid during hysteroscopy procedure
  Arms: Total Capture Drape
Device: Standard Hysteroscopy Drape — Standard surgical drape used to adequately collect fluid during hysteroscopy procedure
  Arms: Control

SUMMARY:
Safety during operative hysteroscopy requires a fluid management system to assist in gauging patient fluid absorption of media used for visualizing the uterine cavity. Serious patient complications, including hyponatremia (low serum sodium), heart failure, and pulmonary and cerebral edema, can result from over absorption of this distending medium. Failure of surgical drapes to collect unabsorbed fluid causes inaccurate determination of the hysteroscopic fluid deficit (HD) thus preventing proper risk evaluation for patient fluid overload, could prompt premature procedure terminatio, and result in hazards for the OR team.

Specific Aims:

1. To perform a comparative trial of the "Total Capture" hysteroscopy drape (TCD) versus the standard drape during patient surgeries to document improved, real-time determination of patient fluid absorption. Pilot testing of a prototype design of the "Total Capture drape" versus the conventional hysteroscopy drape indicated remarkable improvement in fluid capture and accurate fluid deficit determination in a plastic pelvic model experiment.
2. To evaluate the clinical usefulness of the TCD compared to the Standard drape for hysteroscopy with the standardized metrics of: 1) the Technology Acceptance Model, and 2) The System Usability Scale. These metrics will allow us to quantitate clinical usefulness and usability of both the operating surgeons and operating room staff.

The investigators hypothesize the "Total Capture" Drape design provides an accurate recorded hysteroscopic fluid deficit in real-time so that patient safety and surgical parameters are optimized. The simple design of the TCD would add a very significant improvement for patient safety and care with minimal cost for the estimated 200,000 hysteroscopies performed per year in the U.S.

DETAILED DESCRIPTION:
EXPERIMENTAL TRIAL WITH THE TCD VERSUS THE STANDARD HYSTEROSCOPY DRAPE IN A PELVIC MODEL SIMULATION

The investigators sought to document whether or not a prototype design of the "Total Capture" drape (TCD) would perform under replicated clinical conditions in a superior fashion compared to the currently marketed hysteroscopy drape. The experimental testing was performed at an operating room suite using the hysteroscopy fluid management system, conventional hysteroscopy drape, the Total Capture drape and the ZOE Gynecologic pelvic model. The pelvic model was configured so that all fluid introduced into the artificial vagina would not be absorbed by the model but would flow out of the artificial vagina.

A total of four trials per drape were conducted. One trial from each product had procedural difficulties making results invalid.

Results of the Simulation Trial: In four trials of the total capture drape, there was no deficit observed. It was concluded that no major design iterations would be required to move the TCD prototype to the next phase of development

COMPARATIVE TRIAL FOR "PROOF OF CONCEPT" TESTING TO EVALUATE THE EFFICIENCY OF THE TOTAL CAPTURE DRAPE COMPARED TO THE CONVENTIONAL HYSTEROSCOPY DRAPE DURING HYSTEROSCOPIC SURGERY

All women undertaking hysteroscopy are required to have a sterile surgical drape with a fluid capture pouch system to collect the distention media not absorbed by the patient to calculate fluid deficits. Both the TCD and the standard hysteroscopy drape possess the characteristics described above, although design features of the standard drape are deficient. The TCD falls under Class II status, exempt from the 510(k) clearance process in consideration of FDA's approach to similar devices like the standard hysteroscopy drape (Regulation number 21 CRF 878.4370, product code KKX.

The hysteroscopy fluid deficit will be measured by the fluid management system during each hysteroscopy procedure. The uncollected fluid volume seen on the operating room floor and absorbed by the operation blankets and drapes will also be captured, as well as the estimated fluid loss from leaking hysteroscopy joints and gaskets not captured in the collection bag. Procedure time and alarm sounding for exceeding fluid deficit limit will also be recorded.

MEASURES OF DRAPE USABILITY, QUALITY, AND CONVENIENCE

Staff will be asked to complete the System Usability Scale (SUS) to evaluate their perceived clinical usefulness of the TCD and the standard drape. The SUS is a validated 10-item survey for assessing perceived usability that uses a 5-point Likert scale ranging from strongly disagree to strongly agree. To further subjectively and objectively assess the TCD, a human factors and design researcher will observe the surgeries. The human factors researcher will attend the first surgeries to ensure consistent rating with the design researcher who will subsequently observe the remaining surgeries until data saturation is reached. Staff will be asked to speak aloud using the system, which the researcher will record. Further, the researcher will complete an objective human factors assessment tool. These metrics will allow us to quantitate clinical usefulness and usability of both the operating surgeons and operating room staff. These results will not only provide this assessment of the TCD compared to the standard hysteroscopy drape (which is used across ORs within Atrium Health) but will also provide important information to improve the drape if deficiencies are identified.

DATA MANAGEMENT

Case report forms will be developed by the OBGYN clinical research nursing staff in collaboration with Dr. Marshburn and Dr. Zhao. A REDCap database will be created for secure electronic data capture. The data flow will consist of paper data collection for eligibility assessment, baseline data, randomization, operational procedure, fluid measures, surgery outcomes, adverse events, and protocol deviations. The data will be entered into the electronic database within 3 business days of the enrollment.

STATISTICAL METHODS AND SAMPLE SIZE JUSTIFICATION

The primary outcome for the study is the hysteroscopy fluid deficit (HFD) as determined by the fluid management system by subtracting the outflow volume (OV) from the inflow volume (IV) (HFD=IV-OV). Our null hypothesis is Ho: μStandard=μTCD where μ=mean fluid deficit. Our alternative hypothesis is Ho: μStandard>μTCD due to the underestimation of the outflow volume created by the loss of outflow fluid to floors and blankets. If it is assumed the true absorption rates by the patients are the same between the groups due to randomization, by estimating and testing the difference HFD between the two groups a more accurate measure of the uncollected fluid volume (UFV) will be estimated and tested as shown below:

μStandard - μTCD = (μStandard, true absorption + μStandard, UFV) - μTCD, true absorption

* (μ true absorption + μStandard, UFV) - μtrue absorption
* μStandard, UFV The primary analysis for the study will use a general linear model on the HFD with a fixed effect for study group (TCD versus Standard drape) controlling for surgeon and indication for hysteroscopy, the stratification factors for the randomization.

Secondary outcomes include estimated uncollected fluid volume from floor and blankets, occurrence of the fluid deficit alarm sounding, stopping of the operation due to concerns of overabsorption by the patient, and adverse events. Estimated uncollected fluid volume will be analyzed similar to the primary outcome. All other outcomes are categorical and will be compared using Chi-square analyses.

The investigators will sample 10 procedures(or until data saturation) from each arm (TCD vs standard) to conduct qualitative assessments on Usability using the Human Factors Assessment Tool /Acceptance for the for the surgeons and operating team members.For the SUS, the design strategist will collect data on attending physicians only on their first and fifth procedures (the study team may change it to 1st and 3rd if deemed appropriate). The investigators will estimate means or medians with standard deviations (or interquartile ranges) for the items and total scores for the measuresSUS. Both within (1st vs. 5th) and between arms (TCD vs. standard) comparison on total scores of SUS will be conducted. The investigators will compare the two groups using linear mixed models or generalized linear mixed models (depending on the distribution) with a random effect for the procedure to control for correlation of the measures among team members participating in the same procedure.

There is no prior data on HFD in patients to estimate the variability need for the sample size estimation. There is preliminary data from the simulated experiment showing a 100% recovering of loss deficit by the TCD. If it is conservatively assumed the loss deficit will decrease from 40% to 20% of the inflow volume, this would result in a clinically meaningful improvement with an approximate effect size of 0.92 based on the variability of loss deficit in the simulation. Given this, effect size (relative to standard deviation) is used as the primary justification for the number of patients needed for the study. With a sample size of n=34 per arm, there would be 81% power to detect an effect size of 0.7 (0.7*standard deviation of the HFD) with a two sided, two sample t-test (α=0.05). To account for potential missing data of 10%, it is proposed randomizing 76 women (n=38 per arm). With n=34 women in each group, there would also be 80% power to detect an absolute 33% reduction in the proportion of procedures with the alarm sounding due to fluid deficit threshold being reached assuming the proportion in the standard drape arm is 50%. This power was calculated using a Fisher's Exact test for testing proportions between two independent samples. The same power would apply for detecting differences in the proportion of procedures terminated.

DATA SAFETY AND MONITORING

The PI and the study team will meet biweekly to review the study procedures, enrollment (screening and randomization), implementation, protocol deviations, data collection, and adverse events. The biostatistical team will generate monthly reports to monitor screening, enrollment, completeness of data for intervention implementation and outcomes, adverse events, and protocol deviations.

ELIGIBILITY:
Inclusion Criteria:

* Women who are scheduled for a hysteroscopy that require a fluid management system at an Atrium Health operating room facility.

Exclusion Criteria:

* Women will be excluded if they are not acceptable candidates for a hysteroscopy procedure for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Marshburn, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Patients personal health information are confidential. All patient data are de-identified for analysis and reporting

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Capture Drape | Control
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants were all women age 18 and older who were scheduled for an operative hysteroscopy, enrolled and randomized to Total Capture Drape or Control.
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Capture Drape | Control | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.4) | 41.0 (10.5) | 41.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Hysteroscopic Fluid Deficit (HFD) Measured by the Fluid Management System by Subtracting the Outflow Volume (OV) Returned to the Fluid Management System From the Inflow Volume (IV).
Description: Surgery duration, and average of 30 minutes was used to measure hysteroscopic fluid deficit measured by the fulid management system by subtracting the outflow volume returned to the fluid management system from the inflow volume.
Time Frame: Surgery Duration
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Control Group: Control group which used the standard surgical drape used to adequately collect fluid during hysteroscopy procedure
- Total Capture Drape Group: TCD group which used the surgical drape created by Principal Investigator to adequately collect fluid during hysteroscopy procedure
Arm/Group | Control Group | Total Capture Drape Group
Number analyzed (Participants) | 33 | 34
ml | 347.7 (474.1) | 359.1 (606.6)
Statistical Analysis 1: Comparison: Control Group vs Total Capture Drape Group; Test type: Superiority — Power analysis indicated that with a sample size of 34 per arm, would provide 81% power to detect an effect size of 0.7 (0.7*SD of fluid deficit) with a two-sided, two sample t test (a=0.05); p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [-260.7 to 283.4]

2. Secondary Outcome: Number of Participants With Uncollected Distention Fluid Volume Found on Operating Room Floor and Bedding
Description: Uncollected fluid on operating room floor was documented as present or absent.
Time Frame: Surgery Duration
Measure: Count of Participants; unit: Participants
Arm/Group | Total Capture Drape | Control
Number analyzed (Participants) | 34 | 33
Participants | 14 | 21

3. Secondary Outcome: Number of Participants With Hysteroscopy Fluid Management Alarm Activation
Description: Observed if fluid management alarm indicated unsafe level of patient fluid absorption
Time Frame: 1 day (day of procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Total Capture Drape | Control
Number analyzed (Participants) | 34 | 33
Participants | 9 | 4

ADVERSE EVENTS:
Time Frame: Duration of surgery and recovery time which is an average of 90 minutes.
Description: Any adverse events would be reported to the research team and institutional review board.
Arm/Group | Total Capture Drape | Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
We had to stop enrolling due to COVID-19 so the numbers are lower than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT04540952/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04540952/ICF_001.pdf